CLINICAL TRIAL: NCT01806779
Title: Combination Bupropion / Varenicline for Smoking Cessation in Male Smokers
Acronym: ConNic5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Philip Morris USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00042699; 1P50DA027840-01A1 (NIH)
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-10

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; Zyban; Chantix; Nicotine patches; varenicline; bupropion
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chantix (Experimental): For the first 3 days after being switched from Nicotine Replacement Therapy (NRT) (occurring at one week after initiation of nicotine patch treatment, one week before the target Quit Day), smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12-week active treatment duration.
  Interventions: Drug: Chantix; Drug: Nicotine patches
- Chantix + Zyban (Experimental): For the first 3 days after being switched from NRT (occurring at one week after initiation of nicotine patch treatment, one week before the target Quit Day), smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week plus Zyban at a dose of 150mg once per day. Subsequently, the dose of Chantix will be 1 mg twice per day and the dose of Zyban will be 150 mg twice per day for the remainder of the 12-week active treatment duration.
  Interventions: Drug: Chantix; Drug: Zyban; Drug: Nicotine patches

INTERVENTIONS:
Drug: Chantix
  Other Names: Varenicline
Drug: Zyban
  Other Names: Bupropion
  Arms: Chantix + Zyban
Drug: Nicotine patches — All participants will receive 21 mg/24 h dose nicotine (nic.) patches for 1 week.
  Other Names: NRT

SUMMARY:
Previous results from the investigators' Center have shown that combination treatment with Chantix and Zyban is more successful in helping men quit smoking. The investigators hope to replicate these findings with this study.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Male;
* Are 18-65 years old;
* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an expired air carbon monoxide (CO) reading of at least 10ppm;
* Able to read and understand English;
* Express a desire to quit smoking in the next thirty days.

Potential subjects must agree to use acceptable contraception.

Potential subjects must agree to avoid the following:

* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* use of opiate medications.

Exclusion Criteria:

* Hypertension;
* Hypotension with symptoms;
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and electrocardiogram (ECG) clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years;
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease (including but not limited to Chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, Obsessive Compulsive Disorder (OCD) and ADHD);
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression;
* Bulimia or anorexia;
* Use of opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed) within the past 14 days;
* Smoking more than one cigar a month.
* Alcohol abuse;
* Significant adverse reaction to nicotine patches, bupropion / Wellbutrin / Zyban or Chantix / varenicline in the past.
* Current participation or recent participation (in the past 30 days) in another smoking study at our Center or another research facility.
* Current participation in another research study.

Use (within the past 30 days) of:

* Illegal drugs (or if the urine drug screen is positive for tetrahydrocannabinol (THC), Cocaine, Amphetamine, Opiates, Methamphetamines, phencyclidine (PCP), Benzodiazepines, or Barbiturates),
* Experimental (investigational) drugs;
* Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
* Smokeless tobacco (chewing tobacco, snuff), pipes or e-cigarettes;
* Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine replacement therapy or any other smoking cessation aid.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Duke Center for Smoking Cessation, Charlotte, North Carolina
  - Duke Center for Smoking Cessation, Durham, North Carolina
  - Duke Center for Smoking Cessation, Raleigh, North Carolina
  - Duke Center for Smoking Cessation, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Rose JE, Behm FM. Combination Varenicline/Bupropion Treatment Benefits Highly Dependent Smokers in an Adaptive Smoking Cessation Paradigm. Nicotine Tob Res. 2017 Aug 1;19(8):999-1002. doi: 10.1093/ntr/ntw283. PMID 29054128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 3/4/2013 and ended on 9/7/2014. Of the 376 subjects (subjs.) consented during this period, 197 subjects met all study criteria.
Pre-assignment Details: Of the 376 subjs. enrolled, 179 were withdrawn by study staff or withdrew voluntarily from further participation prior to the 1st study visit (V1). 197 subjs. met all study criteria, attended V1 & given NRT for 1 week; 176 subjs. attended V2 & completed SE quest.; 2 subjs. dropped out during this visit before randomization; 174 subjs. randomized.
Groups:
- Chantix: For the first 3 days after being switched from Nicotine Replacement Therapy (NRT, occurring at one week after initiation of nicotine patch treatment, one week before the target Quit Day), smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12-week active treatment duration.
  Chantix
  Nicotine patches: All participants will receive 21 mg/24 h dose nicotine patches for 1 week.
- Chantix + Zyban: For the first 3 days after being switched from NRT (occurring at one week after initiation of nicotine patch treatment, one week before the target Quit Day), smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week plus Zyban at a dose of 150mg once per day. Subsequently, the dose of Chantix will be 1 mg twice per day and the dose of Zyban will be 150 mg twice per day for the remainder of the 12-week active treatment duration.
  Chantix
  Zyban
  Nicotine patches: All participants will receive 21 mg/24 h dose nicotine patches for 1 week.
- Nicotine Patches Only: These subjects received nicotine patches at the first study visit but dropped out before randomization. 176 subjects attended the second study visit and provided side effects (SE) data. Two of these subjects dropped out during that visit (after providing SE data but prior to randomization). So, out of the initial 197 subjects receiving nicotine patches, 174 went on to receive Chantix or Chantix+Zyban; 23 subjects only received nicotine patches before dropping out.
Period: Overall Study
Arm/Group | Chantix | Chantix + Zyban | Nicotine Patches Only
Started | 90 | 84 | 23 (All 197 subjects received nicotine patches but 23 dropped before receiving other study drugs.)
Completed SE Quest. After Using Patches | 90 (SE quest. = Side Effects Questionnaire) | 84 (SE quest. = Side Effects Questionnaire) | 2 (SE quest. = Side Effects Questionnaire)
Randomized at Visit 2 | 90 | 84 | 0
Completed SE Quest. After Randomization | 87 (SE quest. = Side Effects Questionnaire) | 83 (SE quest. = Side Effects Questionnaire) | 0 (SE quest. = Side Effects Questionnaire)
Completed | 48 | 40 | 0
Not Completed | 42 | 44 | 23
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 19 | 20 | 0
Not completed — Withdrawal by Subject | 20 | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chantix | Chantix + Zyban | Total
Number analyzed (Participants) | 90 | 84 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 84 | 174
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.75 (11.381) | 43.12 (10.562) | 43.96 (10.992)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 90 | 84 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 88 | 83 | 171
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 26 | 46
  White | 66 | 57 | 123
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 90 | 84 | 174

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Continuous Four-week Abstinence From Smoking Between the 8-week and 11-week Post Quit Day Visits
Description: This will be determined by a composite of self-report at the 11-week study visit of no smoking between the 8-week and 11-week visits and expired air carbon monoxide (CO) <10 ppm (measured at the 11-week study visit). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.
Time Frame: Period between 8-week and 11-week visits post target Quit Day
Measure: Number; unit: participants
Arm/Group | Chantix | Chantix + Zyban
Number analyzed (Participants) | 90 | 84
participants | 41 | 38

2. Secondary Outcome: Number of Participants Completing Seven-day Point Abstinence From Smoking at 6 Months Post Quit Day
Description: This will be determined by a self-report of no smoking for the previous seven days when called for 6-month follow-up confirmed by expired air CO.
Time Frame: 6 months post Quit Day
Measure: Number; unit: participants
Arm/Group | Chantix | Chantix + Zyban
Number analyzed (Participants) | 90 | 84
participants | 21 | 19

3. Secondary Outcome: Number of Participants Completing Continuous Abstinence From Smoking Between Quit Day and 11-week Post Quit Day Visit
Description: This will be determined by a composite of self-report of no smoking between study visits at the 1-week, 3-week, 7-week and 11-week post Quit Day study visits and expired air carbon monoxide (CO) <10 ppm (measured at those study visits). An intent-to-treat criterion will be used, whereby drop-outs are considered to be non-abstinent.
Time Frame: Quit Day to 11-week post Quit Day study visit
Measure: Number; unit: participants
Arm/Group | Chantix | Chantix + Zyban
Number analyzed (Participants) | 90 | 84
participants | 21 | 15

4. Other Pre Specified Outcome: Change in Smoking Withdrawal Symptoms
Description: Withdrawal symptoms will be assessed by questionnaire on Quit Day, Week 1, Week 3, Week 7 and Week 11 post target quit date and 6 months post quit Follow-Up (if applicable) using the Shiffman-Jarvik questionnaire, which consists of 33-items rated from 1 to 7, where 1= not at all, 2= very little, 3= a little, 4= moderately, 5= a lot, 6= quite a lot, and 7= extremely. The 33 items are grouped into 8 subscales: Craving, Negative Affect, Appetite, Arousal, Somatic - Anxiety, Somatic - G.I., Somatic - Respiratory Tract, and Habit Withdrawal. The range of scores for each subscale will be 1-7, with higher scores indicating more of the withdrawal symptom having been experienced.
Time Frame: Quit Day and 1 week, 3 weeks, 7 Weeks, 11 Weeks and 6 months post Quit Day
Population: A total of 163 subjects (Chantix n=82, Chantix+Zyban n=81) attended the first post-quit visit. However, ten subjects (5 in each condition) failed to complete or return their Quit Day withdrawal questionnaires; therefore change scores could only be calculated for 153 subjects (Chantix n=77, Chantix+Zyban n=76).
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Chantix | Chantix + Zyban
Number analyzed (Participants) | 77 | 76
percentage of change
  Craving -- % change 1 week from Quit Day | -18.15 (2.354) | -15.49 (3.117)
  Craving -- % change 3 weeks from Quit Day | -27.06 (3.520) | -28.64 (4.439)
  Craving -- % change 7 weeks from Quit Day | -30.94 (3.124) | -28.75 (5.104)
  Craving -- % change 11 weeks from Quit Day | -26.97 (4.471) | -30.82 (5.201)
  Craving -- % change 6 months from Quit Day | -42.96 (6.563) | -33.52 (9.020)
  Negative Affect -- % change 1 week from Quit Day | -11.45 (2.551) | -7.15 (2.791)
  Negative Affect -- % change 3 weeks from Quit Day | -9.74 (2.494) | -4.72 (4.230)
  Negative Affect -- % change 7 weeks from Quit Day | -10.16 (2.885) | -10.88 (4.177)
  Negative Affect -- % change 11 weeks from Quit Day | -15.06 (3.396) | -8.52 (4.567)
  Negative Affect -- % change 6 months from Quit Day | -8.55 (10.707) | 21.96 (19.660)
  Appetite -- % change 1 week from Quit Day | -10.53 (3.148) | -4.40 (3.224)
  Appetite -- % change 3 weeks from Quit Day | -11.04 (5.065) | -4.42 (5.553)
  Appetite -- % change 7 weeks from Quit Day | -9.30 (5.981) | -11.66 (6.403)
  Appetite -- % change 11 weeks from Quit Day | -16.20 (7.153) | -8.64 (8.199)
  Appetite -- % change 6 months from Quit Day | -33.88 (10.872) | -35.44 (15.819)
  Arousal -- % change 1 week from Quit Day | 8.03 (5.620) | 10.72 (3.716)
  Arousal -- % change 3 weeks from Quit Day | 5.87 (5.675) | -4.40 (3.643)
  Arousal -- % change 7 weeks from Quit Day | 6.94 (6.763) | -4.03 (3.950)
  Arousal -- % change 11 weeks from Quit Day | 7.33 (6.117) | -1.56 (3.928)
  Arousal -- % change 6 months from Quit Day | 19.80 (15.516) | 49.01 (32.352)
  Anxiety -- % change 1 week from Quit Day | -8.22 (3.480) | -12.26 (2.780)
  Anxiety -- % change 3 weeks from Quit Day | -8.66 (4.001) | -14.40 (3.517)
  Anxiety -- % change 7 weeks from Quit Day | -11.82 (3.25) | -12.50 (5.000)
  Anxiety -- % change 11 weeks from Quit Day | -9.34 (3.526) | -19.83 (3.768)
  Anxiety -- % change 6 months from Quit Day | -66.77 (3.269) | -57.15 (6.064)
  Gastrointestinal -- % change 1 week from Quit Day | -0.69 (3.720) | -7.78 (2.692)
  Gastrointestinal -- % change 3 weeks from Quit Day | -5.14 (2.994) | -10.07 (2.791)
  Gastrointestinal -- % change 7 weeks from Quit Day | -7.67 (3.231) | -8.44 (4.777)
  Gastrointestinal - % change 11 weeks from Quit Day | -8.05 (3.357) | -9.60 (3.897)
  Gastrointestinal - % change 6 months from Quit Day | -67.72 (3.245) | -56.61 (6.026)
  Respiratory -- % change 1 week from Quit Day | 1.41 (3.113) | -7.47 (2.887)
  Respiratory -- % change 3 weeks from Quit Day | -1.12 (4.694) | -8.81 (3.697)
  Respiratory -- % change 7 weeks from Quit Day | 0.92 (6.534) | -18.04 (4.120)
  Respiratory -- % change 11 weeks from Quit Day | -4.36 (6.014) | -19.67 (4.507)
  Respiratory -- % change 6 months from Quit Day | -65.87 (3.293) | -55.77 (6.618)
  Habit -- % change 1 week from Quit Day | -5.15 (4.878) | 1.64 (5.120)
  Habit -- % change 3 weeks from Quit Day | -17.67 (4.959) | -16.07 (3.735)
  Habit -- % change 7 weeks from Quit Day | -14.46 (6.666) | -20.55 (4.868)
  Habit -- % change 11 weeks from Quit Day | -16.61 (6.601) | -24.78 (6.085)
  Habit -- % change 6 months from Quit Day | -56.97 (4.807) | -53.40 (5.905)

ADVERSE EVENTS:
Time Frame: Subjects (subjs.) received (rcvd.) study drugs for 13 weeks. At each study session during this period subjs. completed a questionnaire about side effects (SE). Subjs. were also told to contact study staff between study sessions if SE were bothersome.
Description: Serious Adverse Events (AE) were evaluated for all subjs. who rcvd. nic. patches at Visit (V) 1 (197), & subjs. randomized to receive Chantix (90) or Chantix+Zyban (84) at V2. Other AEs were evaluated for all subjs. receiving nic. patches & completing V2 SE quest. (176), & randomized subjs. completing SE quest. at V3 (170) & at subsequent visits.
Groups:
- Chantix + Zyban: For the first 3 days after being switched from Nicotine Replacement Therapy (NRT, occurring at one week after initiation of nicotine patch treatment, one week before the target Quit Day), smokers in this group will receive treatment with Chantix at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week plus Zyban at a dose of 150mg once per day. Subsequently, the dose of Chantix will be 1 mg twice per day and the dose of Zyban will be 150 mg twice per day for the remainder of the 12-week active treatment duration.
  Chantix
  Zyban
  Nicotine patches: All participants will receive 21 mg/24 h dose nicotine patches for 1 week.
- Nicotine Patch: All participants will receive Nicotine Replacement Therapy (NRT) in the form of 21 mg/24 h dose nicotine patches for 1 week prior to randomization to treatment with Chantix alone or Chantix + Zyban.
Arm/Group | Chantix | Chantix + Zyban | Nicotine Patch
Serious Adverse Events (participants affected / at risk) | 3/90 | 2/84 | 0/197
Other Adverse Events (participants affected / at risk) | 39/87 | 53/83 | 57/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chantix (N=90) | Chantix + Zyban (N=84) | Nicotine Patch (N=197)
Allergic Reaction to Chantix or Zyban (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac Chest Pain & Right Ventricular Hypertrophy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Jaw & upper extremity fracture due to an accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
COPD and reactive airway disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Left sided weakness, headache, blurred vision (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chantix (N=87) | Chantix + Zyban (N=83) | Nicotine Patch (N=176)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3)
Excessive Sweating (Nervous system disorders) | 2 (3) | 7 (11) | 4 (4)
Change in Taste (Nervous system disorders) | 4 (6) | 17 (26) | 4 (4)
Dry Mouth (General disorders) | 8 (13) | 11 (19) | 4 (4)
Thirst (General disorders) | 6 (11) | 15 (32) | 10 (10)
Joint/Muscle/Back Pain (Musculoskeletal and connective tissue disorders) | 4 (10) | 6 (12) | 2 (2)
Irritability (Nervous system disorders) | 8 (12) | 11 (17) | 4 (4)
Vivid Dreams (Nervous system disorders) | 13 (29) | 19 (38) | 30 (30)
Insomnia (Nervous system disorders) | 7 (7) | 8 (17) | 11 (11)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0)
Decreased Libido (General disorders) | 1 (1) | 5 (6) | 2 (2)
Itching/Burning at Patch Site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes